CLINICAL TRIAL: NCT03189368
Title: Heart Failure Study of Multi-site Pacing Effects on Ventriculoarterial Coupling
Acronym: HUMVEE
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Polychronis Dilaveris, Director of Cardiology, First Department of Cardiology, Hippokrateion General Hospital, National and Kapodistrian University of Athens
Other Study IDs: HippoCT1
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Multi-site Pacing; Ventriculoarterial Coupling; Energy Efficiency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Heart failure patients eligible for CRT: Adult, consenting patients with any cardiomyopathy type and an existing I/IIa indication for a CRT-D device will receive a device with multi-site pacing capability. Initially, for 6 months, optimal, conventional, resynchronization therapy will be delivered. Following this, all patients will crossover to optimized multi-site pacing, and receive this therapy for 6 more months. Optimization of therapy will be determined based on maximization of cardiac output, i.e. maximization of left ventricular outflow tract velocity-time integral.
  Baseline measurements of serum creatinine and ventriculoarterial coupling will also be acquired.
  Interventions: Device: Activation of multi-site pacing capability on CRT devices

INTERVENTIONS:
Device: Activation of multi-site pacing capability on CRT devices — Instead of administering a single LV pulse at the most (electrically) delayed segment of the ventricle, multi-site pacing allows for a more detailed "sculpting" of the LV activation sequence. Based on the MPP-IDE study results, activation of the antero-lateral wall, or at least its most delayed segments, closely followed by a pulse to the apex and then by a right ventricular one will yield favorable results in terms of hemodynamics and clinical parameters.
  Programming features:
  * Interpolar distance for the first left ventricular pulse >30mm (i.e. non-sequential poles used)
  * Nearly simultaneous (Δt=5msec) second left ventricular pulse and
  * Threshold of ≤3.5V@0.5msec

SUMMARY:
To perform a comparative study of multi-site left ventricular pacing and cardiac resynchronization therapy effects on ventriculoarterial coupling and energy efficiency of the failing heart

DETAILED DESCRIPTION:
Given that the main function of the cardiovascular system is to provide sufficient blood supply to tissues in order to ensure their normal and effective function, combined with the most efficient possible use of energy produced by ATP degradation, there has been a keen interest in elucidating the interplay between heart and vessels, critically affecting both.

In order to achieve these goals, it is thought that in healthy humans the cardiovascular system as a unity operates at a unique combination of parameters (arterial elastance, heart rate and left ventricular end systolic elastance) so as to:

1. Maximize stroke work (SW) for a given left ventricular contractility. This is related to the fact that adequate tissue perfusion is dependent both on stroke volume and on pressure and in fluid dynamics W=∆P×∆V (thus maximizing SW leads to optimal perfusion), OR
2. Optimize energy efficiency of the heart, in terms of energy transferred to the arterial bed to total mechanical energy.

Ventriculoarterial coupling (VAC) is a composite parameter, defined as the ratio of arterial elastance (Ea) to end systolic left ventricular elastance (Ees). Thus: VAC=Ea/Ees . It is a fundamental property of the cardiovascular system, integrating and assessing the interaction of all individual parameters of the ventricle (pump) and the arterial tree (afterload). Furthermore, VAC may assess both whether SW produced is maximal for a given contractility of the left ventricle (condition for maximization: VAC=1) and whether mechanical efficiency of the ventricle is optimal (optimization condition: VAC=0.5-0.7). Consequently, simultaneous optimization is not possible, and the cardiovascular system operates either at maximal output (as in healthy individuals at rest) or at optimal efficiency (healthy individuals at exercise). Multi-site pacing (MSP) of the left ventricle is a recently introduced technique with excellent studies' findings concerning echocardiographic parameters of ventricular function. Recently, the MultiPoint Pacing (MPP) IDE study showed that a specific choice of electrical dipole for the first left ventricular pulse and a close to simultaneous application of the two left ventricular pulses achieves a very high percent of clinical response (87%), with excellent patient safety. Subsequent studies confirmed these findings, reporting even higher NYHA response rates (95% vs 78% for conventional cardiac resynchronization therapy - CRT).

The underlying rationale lies in the better approximation of the normal sequence of left ventricular activation, through use of two, instead of a single, pulses. According to trial results, one can achieve, compared to conventional CRT, improved coordination between left ventricular segments, improved cardiac output and, possibly, tissue perfusion, and potentially reduction of arrhythmia propensity (mechanism similar to that of CRT). Thus, it would be interesting to study whether these can be independently confirmed by changes in VAC values. In heart failure, VAC values increase considerably due to increases in Ea as a result of the feedback loop regarding pressure (but not volume) maintenance. As a consequence, any reduction would move them closed to both 1 and the 0.5-0.7 area, yielding improvement in both SW maximization and efficiency optimization.

However, there are objective difficulties in achieving lege artis MSP (according to MPP-IDE study standards) given that two prerequisites must be met: 1. Interpolar distance for the first left ventricular pulse >30mm (i.e. non-sequential poles used), 2. Nearly simultaneous (Δt=5msec) left ventricular pulses and 3. Threshold of ≤3.5V@0.5msec.

Moreover, the first pulse should, ideally, be directed to the most delayed, compared to the normal activation sequence, viable myocardial segment, a feat not always possible due to electrode placing constraints. Obviously, presence of scar could alter the course and shape of the activation front and thus diminish its effects (similar to issues already discussed in the case of CRT).

Objective:

To perform a comparative study of multi-site left ventricular pacing and cardiac resynchronization therapy effects on ventriculoarterial coupling and energy efficiency of the failing heart

Hypothesis:

VAC values are improved (shift closer to unity/0.5-0.7 area) and work/efficiency increase with patients on MSP as compared to CRT pacing.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years of age), consenting patients
* Any cardiomyopathy type and
* An existing I/IIa indication for a CRT-D device

Exclusion Criteria:

* Those with a class IIb CRT indication
* Those where thresholds of <3.5V@0.5msec cannot be achieved in at least two dipoles of the left pacing electrode
* Those where no dipole with a distance between poles of 30mm can be detected
* Those with >2/4 (moderate to severe - severe) mitral/aortic insufficiency, rendering noninvasive VAC calculation unreliable.
* Finally, contraindication to receiving intravenous paramagnetic contrast (gadolinium) will also constitute grounds for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systolic heart failure with an ejection fraction of 35% or less, at NYHA functional class of II or worse, and a QRS displaying either LBBB morphology and >120msec or non-LBBB morphology and >150msec.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Improvement of ventriculoarterial coupling | 6 months for each intervention (conventional CRT - MPP)
  Ventriculoarterial coupling value shifts closer to 1
Improvement of energy efficiency | 6 months for each intervention (conventional CRT - MPP)
  Energy efficiency improvement will be assessed by means of ventriculoarterial coupling value shifts closer to 0.7

SECONDARY OUTCOMES:
Improvement in renal function | 6 months for each intervention (conventional CRT - MPP)
  Creatinine clearance (Cockcroft-Gault formula) increases
Improvement in percent maximal stroke work | 6 months for each intervention (conventional CRT - MPP)
  Calculated through use of ventriculoarterial coupling

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Cardiology, Hippokration General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chrysohoou C, Dilaveris P, Antoniou CK, Skiadas I, Konstantinou K, Gatzoulis K, Kallikazaros I, Tousoulis D. Heart failure study of multipoint pacing effects on ventriculoarterial coupling: Rationale and design of the HUMVEE trial. Ann Noninvasive Electrocardiol. 2018 May;23(3):e12510. doi: 10.1111/anec.12510. Epub 2017 Oct 15. PMID 29034563